CLINICAL TRIAL: NCT04954300
Title: Investigation on the Dynamic Changes in Air Microbiome in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2021076
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-05

CONDITIONS: Hospital Acquired Infection
Keywords: Microbial Colonization; Environmental Exposure; Microbiome
MeSH Terms: conditions — Cross Infection; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — We collected the air samples in 3 different ICU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- open: open: open ICU
  Interventions: Other: no intervention
- negative: negative: negative-pressure laminar flow ward
  Interventions: Other: no intervention
- positive: positive: laminar flow ward
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
The microbiome of ICU, especially the air microbiome of ICU is not clear. The relationship between the microbiome of ICU and the hospital- acquired infection needs to be clarified. In this study, we try to outline the dynamic changes of microbiome in ICU and give some advice on the prevention of HAI.

ELIGIBILITY:
Inclusion criteria: no patients were enrolled in this study. Exclusion criteria: no patients were enrolled in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No patients were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Community of microbiome in ICU | 1 year and a half
  the dynamic changes of metagenomic/16s sequencing data

CONTACTS AND LOCATIONS:
Overall Officials: Yuxin Leng, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No